CLINICAL TRIAL: NCT02294513
Title: Hearing Intervention for Patients With Early-Stage Alzheimer's Disease: Determining the Benefits for Patients and Family Caregivers
Brief Title: Hearing Instruments in Alzheimer's Disease
Acronym: HIAD
Status: Completed | Type: Observational
Sponsor: Phonak AG, Switzerland (Industry)
Collaborators: University of Toronto (Other); Baycrest Centre for Geriatric Care (Other)
Responsible Party: Sponsor
Other Study IDs: CHPHST101659-03HIAD
Record Dates: First submitted 2014-10-31; First posted 2014-11-19 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Alzheimer Disease; Hearing Loss
Keywords: Alzheimer disease; Dementia; Hearing loss; Correction of hearing impairment; Hearing aids; Communication; Family caregivers; Third-party disability
MeSH Terms: conditions — Alzheimer Disease; Hearing Loss; Dementia; Communication | interventions — Hearing Aids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- AD_HI: This group will consist of participants with Alzheimer's disease who receive treatment (Standard audiologic rehabilitation (incl. HI)) immediately and are followed over a three-month intervention period.
  Interventions: Device: Standard audiologic rehabilitation (incl. HI)
- NC_HI: This group will consist of participants with normal cognition (i.e., no diagnosis of Alzheimer's disease) who receive treatment (Standard audiologic rehabilitation (incl. HI)) immediately and are followed over a three-month intervention period.
  Interventions: Device: Standard audiologic rehabilitation (incl. HI)

INTERVENTIONS:
Device: Standard audiologic rehabilitation (incl. HI) — The intervention consists of standard audiologic rehabilitation in which participants are fit with at least one hearing instrument (HI).
  Other Names: hearing aid

SUMMARY:
There is a strong connection between hearing loss and cognitive impairment, particularly dementia, in old age. Worldwide, dementia affects approximately 5% of persons over the age of 65 years. Hearing loss is even more prevalent in old age, affecting an estimated one third of persons over the age of 65 years. Thus, there is likely a large degree of overlap between the impairments. Indeed, this overlap may influence older adults' everyday functioning, communication, social engagement and quality of life, as well as influencing the well-being of their family caregivers. This project will examine whether patients with hearing loss and Alzheimer's disease, the most common form of dementia, derive benefit the from hearing aids prescribed and fit to them following current best practice procedures in a geriatric audiology clinic. For the first time, a formal evaluation of the potential benefits of hearing aids for the patients' family caregivers will also be conducted.

DETAILED DESCRIPTION:
Currently, five percent of individuals over the age of 65 suffer from Alzheimer's disease (AD) or a related dementia. Given that hearing loss affects approximately one third of individuals over the age of 65, it is likely that many persons with AD will also suffer from co-morbid hearing loss. Following this logic, a small proportion of the patients treated in a geriatric audiology clinic most likely have both AD and hearing loss. Little research has examined the use of hearing aids by persons with AD, and whether current audiologic rehabilitation can provide benefits for their cognitive, social, and communication functioning. In addition, given that caregiver burden is a huge issue for caregivers of persons with AD, this study will examine whether providing hearing aids to those with AD has concomitant benefits for their family caregivers (e.g., spouse, adult child).

The main research question in this study is: Will persons with AD demonstrate benefit from the use of hearing aids, where benefit is measured through questionnaires assessing activities of daily living, communication, and social functioning. We hypothesize that participants with AD in the intervention group (i.e., those who receive hearing aids) will have a larger improvement in overall functioning at the end of a one-month and three-month period than participants with AD in two control groups. Furthermore, we hypothesize that a group of cognitively normal control participants will demonstrate similar gains in functioning to those participants with AD. Finally, we hypothesize that a similar disparity in benefit between the intervention and control groups will be seen for the participants' caregivers. The specific objectives for this project are to determine, for people with AD if … a) they can benefit from hearing aids based on common audiologic outcome measures, as well as measures of communication function and activities of daily living, and if such benefits depend on variations in current audiologic practice; b) they can benefit from hearing aids with regard to measures of severity of cognitive, behavioural and psychological symptoms of dementia and related caregiver burden; c) hearing aids can bolster their family caregivers' psychological well-being, relationship with, and perceived burden related to caring for and communicating with someone who suffers from both AD and hearing loss, and if specific issues related to communication and audiologic rehabilitation are identified as important by caregivers; and d) the beneficial effects of the hearing aid intervention on the person and their caregiver can be maintained at three months post-fitting.

A randomized control design will be used with three groups of AD patients randomly assigned to 1) intervention (immediate hearing aid fitting), 2) wait-list control (no hearing aid intervention) or 3) active control (no hearing aid intervention + using a new form of fitness technology). A final group of controls with normal cognition will also be tested. All participants will undergo an assessment of their cognition. They and their family caregivers will complete a battery of measures on at least three occasions: once right before the hearing aid fitting is completed to provide a baseline (1), as well as one-month (2) and three-months (3) post-fitting. Participants in the control groups will also complete a set of additional assessments corresponding to the timeline for the hearing aid fitting of participants in the interventions groups (i.e., they will complete 5 assessments rather than 3). In addition to the study sessions, all participants will also complete standard audiology appointments including hearing testing, hearing aid evaluation, hearing aid fitting, and hearing aid checking.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the Audiology department by a physician with a confirmed diagnosis of Alzheimer's disease (or no diagnosis of AD if a normal cognition participant)
* Pure-tone threshold at 3 kHz in excess of 35 dB HL in the worse ear
* 60 years of age or older
* Able to read and communicate well in English
* Allow the researchers access to their medication list throughout the study to assess any changes in medications
* Willing to use one or more hearing aid(s) on a regular basis
* Has a caregiver who…

  * Is a family member
  * Is over the age of 18
  * Is able to read and communicate well in English.
  * Accompanies participant to Baycrest for all necessary appointments
  * Provides qualitative and quantitative assessments of the participant's everyday behaviours and functioning
  * Is willing to learn and support the participant in using hearing aid(s), provide information on their own well-being and communication function
  * If they currently use one or more hearing aid(s), have acquired said aid(s) at least one year prior and are using it/them in a stable fashion.

Exclusion Criteria:

* Suffered a traumatic brain injury or stroke within the past five years
* Has a history of untreated psychiatric illness
* Has an uncorrected deficit in visual acuity or an untreated visual medical issue (e.g., glaucoma, macular degeneration, diabetic retinopathy)
* Suffers from a neurological disorder (e.g., multiple sclerosis, epilepsy)
* Has any untreated medical conditions that could jeopardize participation in the study
* Has been taking medication for their cognitive impairment (e.g., cholinesterase inhibitor, NMDA receptor antagonists) for less than one month.
* Has a caregiver who…

  * Is not cognitively stable (e.g., has been diagnosed with mild cognitive impairment or dementia)
  * Has a terminal medical or untreated psychiatric conditions that could jeopardize their participation in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clients of geriatric hospital and residential living
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Client Oriented Scale of Improvement (COSI): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of communication situations where the participant experiences difficulty (e.g., at church, in a noisy restaurant). Charts change in difficulty over time
Hearing Handicap Inventory of the Elderly (HHIE): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of hearing and communication handicap
International Outcome Inventory for Hearing Aids (IOI-HA): Change over 2months | 1st, 3rd month for AD_HI & NC_HI (4th, 6th month for controls AD_WaitC & AD_ActC resp.)
  Measure of the effectiveness of hearing aid treatments
Self-Assessment of Communication (SAC): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of difficulties caused by an individual's hearing los
Satisfaction with Amplification in Daily Life (SADL): Change over 2months | 1st, 3rd month for AD_HI & NC_HI (4th, 6th month for controls AD_WaitC & AD_ActC resp.)
  Measure of satisfaction with using hearing aids
Significant Other Assessment of Communication (SOAC): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Completed by significant other, measure of a communication partner's hearing difficulties
Significant Other Scale for Hearing Disability (SOS-Hear): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of third-party disability experienced by spouses of older people with hearing impairment

SECONDARY OUTCOMES:
Words-in-noise test (WIN): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Determines the signal-to-noise (SNR) threshold at which the person can correctly recognize 50% of the target words
Dichotic digits test (DDT): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of central auditory processing
Montreal Cognitive Assessment (MoCA): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of cognitive status
Hopkins Verbal-Learning Test (HVLT): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of verbal memory
Brief Visuospatial Memory Test-R (BVMT): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of visual memory
Behavioural Pathology in Alzheimer's disease (BEHAVE-AD): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of problem behaviours demonstrated by individuals with dementia
Neuropsychiatric Inventory Brief (NPI-Q): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of 12 neuropsychiatric symptoms commonly experienced by individuals with dementia
Positive and Negative Affect Schedule (PANAS): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of mood assessing frequency of 10 positive and 10 negative emotions
Geriatric Depression Scale- Short Form (GDS-S): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of depression in older adults
Bristol Activities of Daily Living Scale: Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of instrumental and basic activities of daily living over the past two weeks
Activity and Social Participation Assessment: Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of the frequency of specific activities
Quality of Life in Alzheimer's disease: Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of the domains of physical health, energy, mood, living situation, memory, family, marriage, friends, chores, fun, money, self, and life as a whole
Practical Hearing Test- Revised: Change over 2months | 1st, 3rd month for AD_HI & NC_HI (4th, 6th month for controls AD_WaitC & AD_ActC resp.)
  Measure of objective ability to use hearing aids
Measure of Audiologic Rehabilitation Self-Efficacy for Hearing Aids: Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of ability to use and maintain hearing aid
Perception of Conversation Index- Dementia of the Alzheimer Type: Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of caregivers' strategies for overcoming conversation difficulties
Relationship Satisfaction Questionnaire (RAS): Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of satisfaction with primary relationship
Social Support Questionnaire: Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of level of social support
Zarit Burden Interview- Short Form: Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of burden associated with behavioural impairments and the situation at home
Short-Form Health Survey-12 items: Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of functional health and well-being
Hours of hearing aid use: Change over 3months | 0, 1st, 3rd month (plus 4th and 6th month for controls AD_WaitC & AD_ActC)
  Measure of how many hours the participant is wearing their hearing aid daily

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Pichora-Fuller, Prof., Principal Investigator — University of Toronto
Locations (1):
- Baycrest Center of Geriatric Care, Toronto, Ontario, Canada